CLINICAL TRIAL: NCT03477890
Title: Angina in Patients Without Obstructive Coronary Disease As Revealed by CT Coronary Angiography (Cor-CTCA): an Observational Cohort Study Involving Coronary Function Tests and a Nested Randomised Trial
Brief Title: Coronary Microvascular Function and CT Coronary Angiography (CorCTCA)
Acronym: CorCTCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); British Heart Foundation (Other); Chief Scientist Office of the Scottish Government (Other Government); NHS Greater Clyde and Glasgow (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17/CARD/25
Record Dates: First submitted 2017-10-06; First posted 2018-03-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Angina, Stable; Angina Pectoris, Variant; Microvascular Angina
MeSH Terms: conditions — Angina, Stable; Angina Pectoris, Variant; Microvascular Angina

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, prospective
Who Masked: Participant
Masking Description: Participants are randomised to a 'Disclosed group' (Intervention group) or a 'Not disclosed group' (Standard Care). In the standard care group, coronary function parameters are measured but the results are not disclosed to the attending clinician or the participant. Coronary function is measured in all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (coronary function test results disclosed) (Active Comparator): Coronary function tests are measured and disclosed to the clinician for re-evaluation of the initial diagnosis and treatment as compared with initial angiography. The intervention involves measurement of FFR, CFR, IMR and RRR in a major coronary artery followed by reactivity testing using incremental doses of acetylcholine (10-4 Molar (M), 10-5 M, 10-6 M) to assess endothelial function, bolus of ACh (10-4 M; 100 micrograms) for vasospasm, followed by glyceryl trinitrate (300 micrograms). FFR will be measured in all arteries with a diameter >=2.5 mm and a stenosis 40% to 90% in severity. Endotypes are based on criteria for abnormal coronary vasodilator function, vasospasm and microvascular resistance. The endotypes (diagnostic strata) are: obstructive CAD, vasospastic angina, microvascular angina, mixed (ie both vasospastic and microvascular disorders), endothelial dysfunction (no angina), normal (non-cardiac). A diagnosis may be ruled-in or ruled-out based on the test results.
  Interventions: Diagnostic Test: Stratified medicine involving a diagnostic intervention
- Usual care group (coronary function results not disclosed) (Sham Comparator): Coronary function tests are measured but not disclosed to the attending clinician or the participant. The same coronary function tests are undertaken as in the intervention group. Masking is achieved by obscuring the catheter laboratory monitors from the attending clinician and participant. The effectiveness of masking and protocol adherence is prospectively monitored.
  Interventions: Diagnostic Test: Stratified medicine involving a diagnostic intervention

INTERVENTIONS:
Diagnostic Test: Stratified medicine involving a diagnostic intervention — Adjunctive tests of coronary artery lesion severity (fractional flow reserve) and function at the time of invasive coronary angiography. Diagnostic groups: stable coronary syndromes in patients with obstructive coronary artery disease (mis-classified by non-invasive CTCA) or no-obstructive coronary disease including the following sub-groups (coronary artery vasospasm, microvascular spasm, impaired vasorelaxation due to (1) endothelial dysfunction and/or (2) non-endothelial dysfunction, or unaffected (normal test results).
  Medical management is linked to contemporary clinical guidelines for the management of patients with stable coronary artery disease (European Society of Cardiology (2013), Scottish Intercollegiate Guideline Network (SIGN), 2017).
  Other Names: Adjunctive tests of coronary disease severity and function (disclosed)
  Arms: Intervention group (coronary function test results disclosed)
Diagnostic Test: Stratified medicine involving a diagnostic intervention — Adjunctive tests of coronary artery lesion severity (fractional flow reserve) and function at the time of invasive coronary angiography. Diagnostic groups: stable coronary syndromes in patients with obstructive coronary artery disease (mis-classified by non-invasive CTCA) or non-obstructive coronary disease including the following sub-groups (coronary artery vasospasm, microvascular spasm, impaired vasorelaxation due to (1) endothelial dysfunction and/or (2) non-endothelial dysfunction, or unaffected (normal test results).
  Medical management is linked to contemporary clinical guidelines for the management of patients with stable coronary artery disease (European Society of Cardiology (2013), Scottish Intercollegiate Guideline Network (SIGN), 2017).
  Other Names: Adjunctive tests of coronary disease severity and function (not disclosed, sham control)
  Arms: Usual care group (coronary function results not disclosed)

SUMMARY:
Angina in patients without obstructive coronary artery disease (CAD) is a clinical conundrum and patient management is heterogeneous. Hypothesis: Abnormal coronary function is common and clinically relevant in this population. Design: An observational cohort study and nested randomised controlled diagnostic strategy trial. Methods: 250 patients with known or suspected angina informed by validated questionnaires but without obstructive CAD (<70% stenosis) in an artery >=2.5 mm or structural heart disease, as revealed by CT coronary angiography (CTCA), will be invited to undergo coronary function testing (FFR, CFR, IMR; intra-coronary ACh) during invasive angiography. Patients will be randomised following angiography but before testing coronary function to disclosure of the coronary function test results or not. Treatment decisions by the attending cardiologist will be recorded before and after disclosure of results. Outcomes: Primary: The between-group difference in the reclassification rate of the initial diagnosis using logistic regression, adjusted for baseline factors associated with the likelihood of reclassification of the initial diagnosis. Secondary: Prevalence of microvascular or vasospastic angina; health status reflected by the EuroQol group 5-Dimensions (EQ-5D), Seattle Angina Questionnaire, Illness perception, treatment satisfaction questionnaires and functional status questionnaires; angina medication and adherence. Value: This research will provide new insights into the conundrum of angina in patients without obstructive CAD or structural heart disease.

DETAILED DESCRIPTION:
According to information provided by the British Heart Foundation, there are approximately 2.3 million men and women living with angina in the United Kingdom (UK). In 2014, there were ~247,363 coronary angiograms performed, mostly for the investigation of known or suspected angina, but only about half of the patients have obstructive coronary artery disease (CAD) identified by the angiogram. Considering CT coronary angiography (CTCA), <=1 in 4 patients referred to the Chest Pain Clinic with chest pain of suspected cardiac origin have obstructive CAD identified by the CTCA scan. The explanation for the cause(s) of the chest pain are often unclear, which can be frustrating to patients and clinicians. Small vessel disease, i.e. microvascular or vasospastic angina may be one explanation.

Anatomical imaging of the coronary arteries non-invasively by CTCA or invasively is an insensitive approach for the assessment of coronary function, and even visual assessment of the angiogram for obstructive CAD by invasive angiography or CTCA, may sometimes lead to mis-diagnosis and sub-optimal outcomes. Novel adjunctive tests of coronary function may have incremental diagnostic value to further inform medical decisions. Taken together, the literature and practice guidelines suggest a clinical problem of unmet need, with the potential for benefits to patients and healthcare providers if the diagnostic management can be improved. Our proposal addresses the evidence gap, by exploiting advances in diagnostic tests to gather information on the prevalence of microvascular and vasospastic disorders in patients with angina in whom obstructive CAD has been ruled out. By implementing a diagnostic management strategy in the context of a randomised, blinded, controlled trial, the investigators aim to determine whether use of coronary function tests in relevant patients might be beneficial.

Angina in patients without obstructive CAD and insights from contemporary clinical trials: The Fractional Flow Reserve versus Angiography for Multivessel Evaluation 2 (FAME-2), Scottish COmputed Tomography of the HEART (SCOT-HEART), Prospective Multicenter Imaging Study for Evaluation of Chest Pain (PROMISE), and Clinical Evaluation of Magnetic Resonance Imaging in Coronary Heart Disease 2 (CE-MARC 2) 2 trials focused on the diagnosis and treatment of angina due to obstructive CAD. Paradoxically, the findings in these trials have diagnosed considerable numbers of patients with angina without obstructive CAD. In FAME-2, of 1220 patients with stable CAD, 332 (27%) had non-flow limiting (FFR>0.80) CAD. The distribution of the Canadian Cardiovascular Society angina classes was similar between the randomised patients and those in the registry (p=0.64), as was the prevalence of silent ischaemia (16%; p=0.96). The registry patients were treated with medical therapy and the MACE rate was 9% at 2 years.

In SCOT-HEART, of 4146 patients with suspected angina assessed at the Chest Pain Clinic, 2450 (59%) had confirmed angina (typical or atypical), yet considering the prevalence of obstructive CAD as revealed by CTCA (>70% stenosis in ≥1 major branches or 50% in the left main stem), just 25% had obstructive CAD. In the PROMISE trial, 10,003 participants (n=8939 (89.4%) with typical or atypical angina) were randomised to a strategy of initial anatomical testing with CTCA or to a strategy of functional testing (exercise ECG or stress imaging). Using similar diagnostic criteria as in SCOT-HEART, only 517 (10.7%) of the 4996 participants in the CTCA group had a 'positive' result. No further data were provided to explain the aetiology of the angina in the patients without obstructive CAD.

Most recently, the CE-MARC 2 trial compared diagnostic strategies in patients referred to the Chest Pain Clinic with a pre-test likelihood of CAD of 10% to 90%. All (n=1202) of the participants had a history of angina, with 401 (33.4%) having typical angina. Only a minority of participants had a positive non-invasive test (12.4% in the CMR group, 18.2% in the myocardial perfusion scintigraphy (MPS) group and 13.4% in the NICE Guideline group). Invasive coronary angiography was performed within 12 months of randomisation in 265 (22%) patients. The primary outcome of unnecessary angiography (defined as an FFR>0.8 or quantitative coronary analysis showing no stenosis ≥70% in 1 view or ≥50% in 2 orthogonal views in all coronary vessels ≥2.5 mm diameter), occurred in 139 subjects (12%): 7.5% in the CMR group, 7.1% in the MPS group and 28.8% of participants in the NICE guidelines group. CEMARC 2 was a pragmatic trial and since invasive angiography was not performed in all of the subjects, the causes of the angina in patients with 'negative' non-invasive imaging tests were unclear. Finally, the ISCHEMIA trial investigators have observed that some of the participants enrolled with moderate-severe myocardial ischemia on stress testing (% left ventricular (LV) mass) do not have obstructive CAD. The Changes in Ischemia and Angina over One year among ISCHEMIA trial screen failures with no obstructive coronary artery disease on coronary CT angiography (CIAO-ISCHEMIA) study has been instigated to investigate these patients in greater detail.

In the SCOT-HEART trial, symptoms and quality of life assessed at baseline and 6 months improved less in patients assigned to the CTCA-guided strategy as compared to standard care. This analysis refuted the hypothesis that symptoms and quality of life would improve with a CTCA-guided strategy and it conflicts with the NICE-95 guideline recommendations. Patients in the CTCA group with a change in diagnosis confirming obstructive CAD or excluding CAD had the greatest improvement in symptoms. By contrast, patients with non-obstructive CAD had the least improvement in symptoms. There could be several reasons to explain this finding. Firstly, patient satisfaction may be greater with a definitive diagnosis and treatment plan i.e. 1) normal coronaries - stop treatment, 2) obstructive CAD - percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG), while a result of intermediate CAD with no change in treatment may result in lower patient satisfaction. Secondly, a false negative CTCA result may have occurred in some patients with flow limiting CAD (since objective assessments of flow limiting CAD and/or ischaemia were not performed). Finally, some patients with non-obstructive CAD may have had microvascular disease. Since clinicians may have stopped angina treatment in patients without obstructive CAD, the symptoms of patients who had microvascular angina (and a negative CTCA scan) may have deteriorated.

The design of our study includes a multicentre, observational study involving novel diagnostic tests of coronary function in order to provide information on the prevalence of microvascular and/or vasospastic disease in patients with angina but non obstructive CAD as revealed by CTCA. The CTCA protocol will be undertaken according optimal standards i.e. heart rate control with beta-blocker medication, administration of sublingual nitrate before the CTCA scan, etc. The clinical relevance of additional tests of coronary function will be assessed through a nested randomised strategy trial of management (diagnosis and treatment) guided by the coronary function test results versus standard care guided by angiography. The possibility of occasional CAD misclassification by CTCA (i.e. false negative, obstructive CAD) will also be assessed. Follow-up will include assessments of health, well-being and treatment satisfaction. The wider adoption of anatomical imaging with CTCA as a first-line diagnostic test for the assessment of stable chest pain (NICE-95 guideline update, November 2016), supports the rationale for this research.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of angina or angina-equivalent informed by the Rose Angina questionnaire.
2. Intermediate or no obstructive coronary disease i.e. no coronary stenosis >70% in an artery >2.5 mm, as revealed by CT coronary angiography.

Exclusion Criteria:

1. A health problem that would explain the angina, e.g. anaemia, moderate-severe aortic stenosis, hypertrophic obstructive cardiomyopathy
2. Obstructive disease evident in a coronary artery (diameter >2.5 mm), i.e. >50 - 70% circumferential plaque extending for ≥2 coronary segments, or a stenosis>70% as revealed by CT coronary angiography
3. Lack of informed consent.

   Exclusion from randomisation in the catheter laboratory:
4. Flow-limiting coronary disease defined by a fractional flow reserve (FFR) ≤0.80 in an artery>2.5 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
Final diagnosis | Day 1
  The between-group difference in the reclassification rate of the initial diagnosis based on CTCA vs. final diagnosis after the invasive procedure involving coronary function tests in a a major coronary artery using logistic regression, adjusted for baseline factors associated with the likelihood of reclassification of the initial diagnosis.

SECONDARY OUTCOMES:
Occurrence of abnormal coronary function in a major epicardial coronary artery | Day 1
  To determine the prevalence of microvascular and/or vasospastic angina at the end of the invasive diagnostic procedure (including the coronary angiogram and coronary function tests) in the study population defined as having non obstructive artery disease (CAD) or none as revealed by a CT coronary angiogram for the investigation of known or suspected CAD.
Presence of an obstructive or flow-limiting stenosis in a major coronary artery. | Day 1
  Assess the prevalence of obstructive CAD (e.g. FFR≤0.80) at the time of invasive coronary angiography.
Procedure-related serious adverse events | Day 1
  Safety as reflected by the occurrence of procedure-related serious adverse events
Prevalence of endotypes | Day 1
  Diagnosis of endotypes (disease strata): obstructive CAD, coronary vasospastic angina, microvascular angina, endothelial dysfunction (no angina), normal (non-cardiac, normal coronary function results, no angina).
Cardiovascular risk | Day 1
  Assess the cardiovascular risk of the participants at baseline, as reflected by the validated JBS3 risk score http://www.jbs3risk.com/
Anxiety and depression | Through study completion, 3 years
  Assess the participants' self-reported levels of anxiety and depression using the Patient Health Questionnaire-4, a 4 item inventory rated on a 4 point Likert-type scale (0-3 per item, with a maximum reported score of 6 for anxiety and 6 for depression).
Treatment satisfaction | Through study completion, 3 years
  Assess the participants' self-reported levels of treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM) (scale categories, 2 to 7; a higher response reflects higher treatment satisfaction).
Illness perception | Through study completion, 3 years
  Assess the participants' perception of their illness using the Brief Illness Perception Questionnaire, a 9 item scale reflecting the cognitive and emotional representations of illness. Each item is analysed individually.
Health status EQ-5D | Through study completion, 3 years
  Assess the participants' general health status and self reported quality of life using the EQ5D questionnaire. Health status is measured in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (each is scored on a scale of 1 to 5, with a score of 5 representing the most severe problems or limitations). The visual analog scale ranges from 0 to 100 units, with higher values representing a better outcome.
Health status (Seattle Angina Score) | Through study completion, 3 years
  Health status and symptoms will be assessed at baseline and again at 6 months, 12 months and closeout using the Seattle Angina Questionnaire. The secondary outcome is the within-subject change in Seattle Angina Score score over time.
Functional status | Through study completion, 3 years
  To assess functional status and activity levels as reflected by the Duke Activity Status Index (DASI) at baseline and during follow-up.
Health economics | 36 months
  Assess resource utilisation including primary and secondary care costs for tests, procedures and outpatient visits, and medicines, between the randomised groups
Serum troponin concentration | Through study completion, 3 years
  Assess associations between circulating concentrations of troponin I protein (ng/L) that may be implicated in the pathophysiology of disorders of coronary function.
Physical activity | Through study completion, 3 years
  To assess physical activity levels as reflected by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) with units of activity expressed in minutes/week at baseline and during follow-up. Patients are classified as inactive, moderately active, or HEPA (health-enhancing physical activity) active, depending on how much vigorous/moderate/light exercise they do in a week.
Plasma endothelin-1 | Through study completion, 3 years
  Assess the circulating concentration of big endothelin-1 (pg/mL) peptide in plasma at sampling time-points, baseline and during follow-up. Big endothelin-1 is the stable pre-cursor of endothelin-1 and big endothelin-1 is more stable than endothelin-1 so the former is intended to be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Katriona Brooksbank, PhD, Study Director — University of Glasgow
Locations (3):
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank, Dunbartonshire
  - Forth Valley Royal Hospital, Larbert, Forth Valley
  - Glasgow Royal Infirmary, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
Data access may be possible pending Sponsor approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At study end
URL: https://www.gla.ac.uk/researchinstitutes/healthwellbeing/research/robertsoncentreforbiostatistics/research/researchsupport/

REFERENCES:
- [Background] Sidik NP, Stanley B, Sykes R, Morrow AJ, Bradley CP, McDermott M, Ford TJ, Roditi G, Hargreaves A, Stobo D, Adams J, Byrne J, Mahrous A, Young R, Carrick D, McGeoch R, Corcoran D, Lang NN, Heggie R, Wu O, McEntegart MB, McConnachie A, Berry C. Invasive Endotyping in Patients With Angina and No Obstructive Coronary Artery Disease: A Randomized Controlled Trial. Circulation. 2024 Jan 2;149(1):7-23. doi: 10.1161/CIRCULATIONAHA.123.064751. Epub 2023 Oct 5. PMID 37795617
- [Background] Berry C. Stable Coronary Syndromes: The Case for Consolidating the Nomenclature of Stable Ischemic Heart Disease. Circulation. 2017 Aug 1;136(5):437-439. doi: 10.1161/CIRCULATIONAHA.117.028991. No abstract available. PMID 28760869
- [Background] Bairey Merz CN, Pepine CJ, Walsh MN, Fleg JL. Ischemia and No Obstructive Coronary Artery Disease (INOCA): Developing Evidence-Based Therapies and Research Agenda for the Next Decade. Circulation. 2017 Mar 14;135(11):1075-1092. doi: 10.1161/CIRCULATIONAHA.116.024534. PMID 28289007
- [Background] Ford TJ, Corcoran D, Berry C. Coronary artery disease: physiology and prognosis. Eur Heart J. 2017 Jul 1;38(25):1990-1992. doi: 10.1093/eurheartj/ehx226. No abstract available. PMID 28549103
- [Background] Williams MC, Hunter A, Shah A, Assi V, Lewis S, Mangion K, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJ, Timmis AD, Newby DE; Scottish COmputed Tomography of the HEART (SCOT-HEART) Trial Investigators. Symptoms and quality of life in patients with suspected angina undergoing CT coronary angiography: a randomised controlled trial. Heart. 2017 Jul;103(13):995-1001. doi: 10.1136/heartjnl-2016-310129. Epub 2017 Feb 28. PMID 28246175
- [Background] SCOT-HEART investigators. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. Lancet. 2015 Jun 13;385(9985):2383-91. doi: 10.1016/S0140-6736(15)60291-4. Epub 2015 Mar 15. PMID 25788230
- [Background] Greenwood JP, Ripley DP, Berry C, McCann GP, Plein S, Bucciarelli-Ducci C, Dall'Armellina E, Prasad A, Bijsterveld P, Foley JR, Mangion K, Sculpher M, Walker S, Everett CC, Cairns DA, Sharples LD, Brown JM; CE-MARC 2 Investigators. Effect of Care Guided by Cardiovascular Magnetic Resonance, Myocardial Perfusion Scintigraphy, or NICE Guidelines on Subsequent Unnecessary Angiography Rates: The CE-MARC 2 Randomized Clinical Trial. JAMA. 2016 Sep 13;316(10):1051-60. doi: 10.1001/jama.2016.12680. PMID 27570866
- [Background] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Background] Beltrame JF, Crea F, Kaski JC, Ogawa H, Ong P, Sechtem U, Shimokawa H, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for vasospastic angina. Eur Heart J. 2017 Sep 1;38(33):2565-2568. doi: 10.1093/eurheartj/ehv351. PMID 26245334
- [Background] Ong P, Athanasiadis A, Sechtem U. Patterns of coronary vasomotor responses to intracoronary acetylcholine provocation. Heart. 2013 Sep;99(17):1288-95. doi: 10.1136/heartjnl-2012-302042. Epub 2013 Feb 26. No abstract available. PMID 23442537
- [Background] Douglas PS, Hoffmann U, Patel MR, Mark DB, Al-Khalidi HR, Cavanaugh B, Cole J, Dolor RJ, Fordyce CB, Huang M, Khan MA, Kosinski AS, Krucoff MW, Malhotra V, Picard MH, Udelson JE, Velazquez EJ, Yow E, Cooper LS, Lee KL; PROMISE Investigators. Outcomes of anatomical versus functional testing for coronary artery disease. N Engl J Med. 2015 Apr 2;372(14):1291-300. doi: 10.1056/NEJMoa1415516. Epub 2015 Mar 14. PMID 25773919
- [Background] Ford TJ, Corcoran D, Berry C. Stable coronary syndromes: pathophysiology, diagnostic advances and therapeutic need. Heart. 2018 Feb;104(4):284-292. doi: 10.1136/heartjnl-2017-311446. Epub 2017 Oct 13. PMID 29030424
- [Background] Sidik NP, McEntegart M, Roditi G, Ford TJ, McDermott M, Morrow A, Byrne J, Adams J, Hargreaves A, Oldroyd KG, Stobo D, Wu O, Messow CM, McConnachie A, Berry C. Rationale and design of the British Heart Foundation (BHF) Coronary Microvascular Function and CT Coronary Angiogram (CorCTCA) study. Am Heart J. 2020 Mar;221:48-59. doi: 10.1016/j.ahj.2019.11.015. Epub 2019 Dec 2. PMID 31911341
- [Background] Ford TJ, Yii E, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, McCartney P, Corcoran D, Collison D, Rush C, Stanley B, McConnachie A, Sattar N, Touyz RM, Oldroyd KG, Berry C. Ischemia and No Obstructive Coronary Artery Disease: Prevalence and Correlates of Coronary Vasomotion Disorders. Circ Cardiovasc Interv. 2019 Dec;12(12):e008126. doi: 10.1161/CIRCINTERVENTIONS.119.008126. Epub 2019 Dec 13. PMID 31833416
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Ford TJ, Berry C. Angina: contemporary diagnosis and management. Heart. 2020 Mar;106(5):387-398. doi: 10.1136/heartjnl-2018-314661. Epub 2020 Feb 12. No abstract available. PMID 32054665